CLINICAL TRIAL: NCT00020579
Title: A Phase I Study of an Oral Histone Deacetylase Inhibitor, MS-275, in Refractory Solid Tumors and Lymphomas
Brief Title: MS-275 in Treating Patients With Advanced Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 010124; 01-C-0124; NCI-2792; CDR0000068615; NCT00012571 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Cancer
Keywords: stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; small intestine lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; primary central nervous system non-Hodgkin lymphoma; intraocular lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; male breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; recurrent pancreatic cancer; stage III pancreatic cancer; recurrent colon cancer; stage III colon cancer; stage IV colon cancer; recurrent rectal cancer; stage III rectal cancer; stage IV rectal cancer; recurrent ovarian epithelial cancer; recurrent ovarian germ cell tumor; stage III ovarian epithelial cancer; stage III ovarian germ cell tumor; stage IV ovarian epithelial cancer; stage IV ovarian germ cell tumor; recurrent malignant testicular germ cell tumor; stage III malignant testicular germ cell tumor; recurrent cervical cancer; stage III cervical cancer; stage IVA cervical cancer; stage IVB cervical cancer; recurrent endometrial carcinoma; stage III endometrial carcinoma; stage IV endometrial carcinoma; fallopian tube cancer; primary peritoneal cavity cancer; recurrent uterine sarcoma; stage III uterine sarcoma; stage IV uterine sarcoma; recurrent vaginal cancer; stage III vaginal cancer; stage IVA vaginal cancer; stage IVB vaginal cancer; recurrent vulvar cancer; stage III vulvar cancer; stage IV vulvar cancer; recurrent anal cancer; stage IIIA anal cancer; stage IIIB anal cancer; stage IV anal cancer; recurrent esophageal cancer; stage III esophageal cancer; stage IV esophageal cancer; recurrent gastric cancer; stage III gastric cancer; stage IV gastric cancer; recurrent extrahepatic bile duct cancer; unresectable extrahepatic bile duct cancer; advanced adult primary liver cancer; localized unresectable adult primary liver cancer; recurrent adult primary liver cancer; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage III verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; recurrent basal cell carcinoma of the lip; recurrent squamous cell carcinoma of the lip and oral cavity; stage III basal cell carcinoma of the lip; stage III squamous cell carcinoma of the lip and oral cavity; stage IV basal cell carcinoma of the lip; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent lymphoepithelioma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage III lymphoepithelioma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage IV lymphoepithelioma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; recurrent lymphoepithelioma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; stage III lymphoepithelioma of the nasopharynx; stage III squamous cell carcinoma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent inverted papilloma of the paranasal sinus and nasal cavity; recurrent midline lethal granuloma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage III inverted papilloma of the paranasal sinus and nasal cavity; stage III midline lethal granuloma of the paranasal sinus and nasal cavity; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage IV inverted papilloma of the paranasal sinus and nasal cavity; stage IV midline lethal granuloma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; metastatic parathyroid cancer; recurrent parathyroid cancer; recurrent salivary gland cancer; stage III salivary gland cancer; stage IV salivary gland cancer; recurrent bladder cancer; recurrent gallbladder cancer; stage III bladder cancer; stage IV bladder cancer; unresectable gallbladder cancer; recurrent renal cell cancer; stage III renal cell cancer; stage IV renal cell cancer; stage III Wilms tumor; stage IV Wilms tumor; stage V Wilms tumor; metastatic transitional cell cancer of the renal pelvis and ureter; recurrent transitional cell cancer of the renal pelvis and ureter; regional transitional cell cancer of the renal pelvis and ureter; anterior urethral cancer; posterior urethral cancer; recurrent urethral cancer; recurrent penile cancer; stage III penile cancer; stage IV penile cancer; recurrent prostate cancer; stage III prostate cancer; stage IV prostate cancer; metastatic Ewing sarcoma/peripheral primitive neuroectodermal tumor; recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor; metastatic osteosarcoma; recurrent osteosarcoma; recurrent adult soft tissue sarcoma; stage III adult soft tissue sarcoma; stage IV adult soft tissue sarcoma; classic Kaposi sarcoma; AIDS-related Kaposi sarcoma; recurrent Kaposi sarcoma; stage III cutaneous T-cell non-Hodgkin lymphoma; ciliary body and choroid melanoma, medium/large size; ciliary body and choroid melanoma, small size; extraocular extension melanoma; iris melanoma; recurrent intraocular melanoma; recurrent melanoma; stage III melanoma; stage IV melanoma; extensive stage small cell lung cancer; recurrent non-small cell lung cancer; recurrent small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent thymoma and thymic carcinoma; advanced malignant mesothelioma; recurrent malignant mesothelioma; recurrent adrenocortical carcinoma; stage III adrenocortical carcinoma; stage IV adrenocortical carcinoma; metastatic gastrointestinal carcinoid tumor; recurrent gastrointestinal carcinoid tumor; regional gastrointestinal carcinoid tumor; desmoid tumor; newly diagnosed carcinoma of unknown primary; recurrent carcinoma of unknown primary; undifferentiated carcinoma of unknown primary; carcinoma of the appendix; recurrent metastatic squamous neck cancer with occult primary; untreated metastatic squamous neck cancer with occult primary; recurrent pituitary tumor; adult anaplastic astrocytoma; adult astrocytic tumors; adult diffuse astrocytoma; adult pilocytic astrocytoma; adult anaplastic oligodendroglioma; adult brain stem glioma; adult oligodendroglioma; adult mixed glioma; adult central nervous system germ cell tumor; adult choroid plexus tumor; adult craniopharyngioma; adult anaplastic ependymoma; adult subependymoma; adult medulloblastoma; adult supratentorial primitive neuroectodermal tumor (PNET); adult ependymoblastoma; adult ependymoma; adult myxopapillary ependymoma; adult anaplastic meningioma; adult meningeal hemangiopericytoma; adult meningioma; adult papillary meningioma; adult grade I meningioma; adult grade II meningioma; adult grade III meningioma; adult pineal parenchymal tumor; recurrent adult brain tumor; stage IV pancreatic cancer; stage III thymoma; stage IVA thymoma; stage IVB thymoma
MeSH Terms: conditions — Neoplasms; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Intraocular Lymphoma; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Mycosis Fungoides; Sezary Syndrome; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Breast Neoplasms, Male; Breast Neoplasms; Pancreatic Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Carcinoma, Ovarian Epithelial; Testicular Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms; Fallopian Tube Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms; Anus Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Bile Duct Neoplasms; Carcinoma, Hepatocellular; Squamous Cell Carcinoma of Head and Neck; Esthesioneuroblastoma, Olfactory; Parathyroid Neoplasms; Salivary Gland Neoplasms; Urinary Bladder Neoplasms; Gallbladder Neoplasms; Carcinoma, Renal Cell; Wilms Tumor; Urethral Neoplasms; Penile Neoplasms; Prostatic Neoplasms; Neuroectodermal Tumors, Primitive, Peripheral; Osteosarcoma; Sarcoma; AIDS-related Kaposi sarcoma; Sarcoma, Kaposi; Uveal Melanoma; Melanoma; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Thymoma; Mesothelioma, Malignant; Adrenocortical Carcinoma; Desmoid Tumors; Neoplasms, Unknown Primary; Appendiceal Neoplasms; Pituitary Neoplasms; Astrocytoma; Oligodendroglioma; Glioma; Choroid Plexus Neoplasms; Craniopharyngioma; Ependymoma; Glioma, Subependymal; Medulloblastoma; Neuroectodermal Tumors, Primitive; Meningioma; Pinealoma; Brain Neoplasms | interventions — entinostat

INTERVENTIONS:
Drug: entinostat

SUMMARY:
RATIONALE: MS-275 may stop the growth of cancer cells by blocking the enzymes necessary for their growth.

PURPOSE: This phase I trial is studying the side effects and best dose of MS-275 in treating patients with advanced solid tumors or lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the dose-limiting toxicity and maximum tolerated dose of MS-275 in patients with advanced solid tumors or lymphomas.
* Determine the profile of adverse events, including changes in laboratory parameters, in patients treated with this drug.
* Assess the pharmacology and pharmacokinetics of this drug in these patients.
* Design MS-275 regimens with possibly more frequent dose administration based on the pharmacology of MS-275 using the schedule in this study.
* Determine the antineoplastic activity of this drug in these patients.

OUTLINE: This is an open-label, dose-escalation study.

Patients receive oral MS-275 once on day 1. Courses repeat every 2 weeks (every 2-week schedule). Alternatively, patients receive oral MS-275 once on days 1, 8, 15, and 22 (weekly schedule). Courses repeat every 6 weeks. Treatment for both schedules continues in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of MS-275 on the every 2-week schedule until the maximum tolerated dose (MTD) is determined. Once the MTD for the every 2-week schedule is determined, patients receive treatment on the weekly schedule as above. The MTD is then determined for the weekly schedule. The MTD for both schedules is defined as the dose preceding that at which at least 2 of up to 6 patients experience dose-limiting toxicity. Once the MTD is determined for the weekly schedule, up to 3 additional patients are accrued to receive MS-275 at the MTD of the weekly schedule.

Disease status is assessed every 3 months.

PROJECTED ACCRUAL: A total of 50-75 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignancy that is metastatic or unresectable and for which no effective standard curative or palliative therapy exists
* Brain metastases allowed provided both of the following criteria are met:

  * Received treatment for the brain metastases
  * Stable for ≥ 6 months without steroids or antiseizure medications

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2 OR
* Karnofsky 50-100%

Life expectancy:

* More than 3 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN) (≤ 3 mg/dL for patients with Gilbert's syndrome)
* AST/ALT no greater than 2.5 times ULN
* Albumin at least 75% of lower limit of normal

Renal:

* Creatinine normal OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* Cardiac ejection fraction normal by MUGA
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Adequate oral intake
* No weight loss of more than 10% of actual body weight within the past 2 months
* No history of allergic reaction to compounds of similar chemical or biological composition to study drug
* No other uncontrolled illness
* No ongoing or active infection
* No seizure disorder
* No psychiatric illness or social situation that would preclude study compliance
* No acute or chronic gastrointestinal conditions (e.g., peptic ulcer or colitis) within the past 2 months that would interfere with drug tolerance or absorption
* Willing and able to self-administer and document doses of MS-275

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior anticancer vaccine therapy and recovered
* No concurrent immunotherapy

Chemotherapy:

* At least 4 weeks since prior anticancer chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* At least 8 weeks since prior UCN-01 and recovered
* No concurrent chemotherapy

Endocrine therapy:

* At least 4 weeks since prior anticancer hormonal therapy (except gonadotropin-releasing hormone [GnRH] agonists) and recovered
* Concurrent corticosteroids for physiological replacement, as antiemetic therapy, or for an ongoing condition allowed

  * Must be on a stable dose during the past 4 weeks
* No concurrent anticancer hormonal therapy except GnRH agonists for noncastrated patients with prostate cancer

Radiotherapy:

* At least 4 weeks since prior anticancer radiotherapy and recovered
* No concurrent radiotherapy

  * Concurrent localized radiotherapy to a single lesion allowed if the patient achieves at least a partial response

Surgery:

* At least 3 weeks since prior major surgery

Other:

* No other concurrent investigational or commercial antineoplastic therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2001-03; Primary Completion 2008-04 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicities and maximum tolerated dose
Pharmacology and pharmacokinetics

SECONDARY OUTCOMES:
Acetylation of histones in peripheral blood
Tumor response by CT scan every 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shivaani Kummar, MD, Principal Investigator — NCI - Medical Oncology Branch
Locations (3):
- United States (3):
  - National Naval Medical Center, Bethesda, Maryland
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - NCI - Center for Cancer Research, Bethesda, Maryland

REFERENCES:
- [Result] Ryan QC, Headlee D, Sparreboom A, et al.: A phase I trial of an oral histone deacetylase inhibitor, MS-275, in advanced solid tumor and lymphoma patients. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-802, 2003.